CLINICAL TRIAL: NCT07397221
Title: The Effect of Oropharyngeal Humidification After Extubation on Thirst, Pain, and Anxiety in Patients Undergoing Coronary Artery Bypass Surgery: A Randomized Controlled Study
Brief Title: Oropharyngeal Humidification After Extubation on Thirst
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, tasci, Ph.D., Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 218984
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Bypass
Keywords: Oropharyngeal Humidification; Thirst; Pain; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oropharyngeal Humidification (Experimental): Participants in this arm will receive oropharyngeal humidification with room-temperature drinking water spray. After tracheal extubation, the researcher applies the spray to multiple oral regions (upper jaw, lower jaw, left cheek, right cheek, tongue) twice per hour for 4 hours.
  Interventions: Other: Oropharyngeal Humidification with Water Spray
- Routine Oral Care (No Intervention): Participants receive only routine oral care provided in the ICU. Nurses use standard methods such as moistening the mouth with wet cotton swabs or lip wetting as needed.

INTERVENTIONS:
Other: Oropharyngeal Humidification with Water Spray — Room-temperature drinking water is administered as an oral spray to multiple areas of the oral cavity (upper jaw, lower jaw, left and right cheek, and tongue). The researcher applies the spray twice per hour for 4 hours after extubation in patients undergoing coronary artery bypass surgery.
  Arms: Oropharyngeal Humidification

SUMMARY:
In patients who have undergone endotracheal intubation following cardiac surgery, symptoms such as thirst, dysphagia (difficulty swallowing), restlessness, nausea, and vomiting are frequently observed, and these conditions negatively affect the patients' overall comfort. Especially in the post-intubation period, dryness in the mouth and throat, an intense feeling of thirst, and difficulty swallowing can lead to feelings of suffocation, helplessness, fear, and anxiety in patients. Effective management of these symptoms is critically important both for accelerating the recovery process and for increasing patient satisfaction.

Traditionally, methods such as moistening the mouth with a cotton swab have been used to relieve complaints like thirst and dry mouth. However, these practices are often insufficient and have limited effectiveness in increasing patients' comfort. In recent years, the use of oropharyngeal sprays has emerged as an innovative and effective approach to alleviate symptoms such as thirst and dry mouth. In a randomized controlled trial conduct, it was shown that a spray-based oropharyngeal moisturizing program significantly reduced the severity of thirst and discomfort in patients who underwent intubation after cardiac surgery. Thirst and discomfort scores were found to be significantly lower in the spray-applied groups compared to the control group, and no significant difference was observed between the groups in terms of dysphagia frequency or adverse events. Similarly, studies conducted in different surgical and intensive care populations have shown that applications of cold water or cold saline sprays significantly reduce complaints of thirst and dry mouth, increase patient comfort, and are safe to use.

Additionally, it has been reported that alternative approaches such as menthol lozenges or aromatherapy also have positive effects on thirst, nausea, and comfort after cardiac surgery. Examining the effects of oropharyngeal sprays and similar practices on parameters such as thirst, dysphagia, discomfort, nausea, vomiting, and overall comfort in patients who are intubated after cardiac surgery may contribute to the development of innovative and effective approaches in patient care. Integrating such practices into postoperative care protocols carries significant potential for increasing patient comfort and supporting the recovery process.

This randomized controlled study aims to investigate the effects of oropharyngeal humidification after extubation on thirst, pain, and anxiety in patients undergoing coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Undergoing coronary artery bypass surgery
* Postoperative mechanical ventilation and extubation
* Able to provide informed consent

Exclusion Criteria:

* Neuromuscular diseases (e.g., stroke, Parkinson's disease)
* Head/neck deformities
* Pre-existing dysphagia
* Tracheostomy
* Inability to participate in assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Thirst Severity | Baseline (immediately after extubation) 2 hours post-intervention 4 hours post-intervention
  The Numeric Rating Scale is used for patients to indicate the severity of their thirst. Patients will be asked to rate their feeling of thirst on a scale from 0 to 10. A score of 0 means no thirst at all. An increase in the score indicates increasing thirst. A score of 10 represents extreme thirst.

SECONDARY OUTCOMES:
Thirst-Related Discomfort | Baseline (immediately after extubation) 2 hours post-intervention 4 hours post-intervention
  The Perioperative Thirst Discomfort Scale is a 3-point Likert-type scale consisting of a total of 7 items. The rating is as follows: Did not disturb (0), Slightly disturbed (1), and Greatly disturbed. The scale does not have any sub-dimensions. Higher scores indicate greater thirst. The total score on the scale ranges from a minimum of 0 to a maximum of 12.
Pain Severity | Baseline (immediately after extubation) 2 hours post-intervention 4 hours post-intervention
  Visual Analog Scale is used to assess pain. The patient's pain is evaluated with a score between 0 and 10. A score of 0 indicates no pain, while a score of 10 represents unbearable pain. An increase from 0 to 10 indicates increasing pain.
Anxiety Level | Baseline (immediately after extubation) 2 hours post-intervention 4 hours post-intervention
  The State Anxiety Scale is a 20-item, 4-point Likert-type scale. The rating is as follows: Almost never (1), Sometimes (2), Often (3), and Almost always (4). As the score increases, anxiety also increases. The minimum total score on the scale is 0, and the maximum is 80.
Post-Extubation Complications | Continuous monitoring during the 4-hour intervention period
  Complications such as coughing, oxygen desaturation, nausea-vomiting, or dysphagia are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Şehit Prof. Dr. İlhan Varank Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] References Lin, R., Chen, H., Chen, L., Lin, X., He, J., & Li, H. (2022). Effects of a spray-based oropharyngeal moisturising programme for patients following endotracheal extubation after cardiac surgery: A randomised, controlled three-arm trial.. International journal of nursing studies, 130, 104214. https://doi.org/10.1016/j.ijnurstu.2022.104214 Gungor, S., Tosun, B., Candir, G., & Ozen, N. (2024). Effects of cold spray on thirst, frequency of oral care, and pain of general surgery intensive care unit patients. Scientific Reports, 14. https://doi.org/10.1038/s41598-024-58199-0 Lian, R., Zhou, S., Guo, Y., Liang, H., Lin, J., Li, D., Wu, W., Rao, Y., Shao, D., Zheng, P., & Yang, X. (2024). The effect of ice-cold water spray following the model for symptom management on postoperative thirst in patients admitted to intensive care unit: A randomized controlled study.. Intensive & critical care nursing, 81, 103571. https://doi.org/10.1016/j.iccn.2023.103571 Wu, H., Chaou, C., Chang, C., & Wang, H. (2024). [The Comparative Effectiveness of Using Cold Water Oral Spray and Cold Saline Oral Spray for Thirst Relief in Patients With Endotracheal Intubation in the Intensive Care Unit].. Hu li za zhi The journal of nursing, 71 3, 33-42. https://doi.org/10.6224/jn.202406_71(3).06 Ghasemi, A., Mazloum, S., Pourghaznein, T., & Eshraghi, A. (2025). The Impact of Cold Spray Use on Thirst Distress, Dry Mouth, and Fluid Intake in Heart Failure Patients: A Randomized Controlled Study.. The Journal of cardiovascular nursing. https://doi.org/10.1097/jcn.0000000000001183 Liang, T., Li, S., Peng, Y., Chen, Q., Chen, L., & Lin, Y. (2022). Efficacy and Safety of Oral Hydration 1 Hour After Extubation of Patients Undergoing Cardiac Surgery. The Journal of Cardiovascular Nursing, 40, E1 - E8. https://doi.org/10.1097/jcn.0000000000000953 Oztaş, M., & Oztas, B. (2022). Effect of Spray Use on Mouth Dryness and Thirst of Patients Undergoing Maj